CLINICAL TRIAL: NCT05985577
Title: Mechanism of Gastric Signet Ring Cell Carcinoma Based on Microproteomics
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Zhejiang Cancer Hospital (Other)
Responsible Party: Principal Investigator, Xiangdong Cheng, Secretary of the party committee, Zhejiang Cancer Hospital
Other Study IDs: IRB-2023-584
Record Dates: First submitted 2023-07-17; First posted 2023-08-14 (Actual); Last update posted 2023-08-14 (Actual); Status verified 2023-08

CONDITIONS: Gastric Cancer; Signet Ring Cell Carcinoma
Keywords: Gastric signet ring cell carcinoma; Molecular Subtypes; Proteomics; Prognostic markers; Drug target
MeSH Terms: conditions — Stomach Neoplasms; Carcinoma, Signet Ring Cell

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Biospecimen Retention: Samples Without DNA — Biological samples are used for proteomic analysis.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cancer tissues: Cancer tissues
  Interventions: Other: Without any intervention
- Normal adjacent tissues: Normal adjacent tissues
  Interventions: Other: Without any intervention

INTERVENTIONS:
Other: Without any intervention — There were no special interventions for the two groups.

SUMMARY:
Gastric signet ring cell carcinoma (GSRCC) possesses unique epidemiology and pathogenesis in the field of cancer, but its incidence is low. Unfortunately, there is currently a lack of systematic research focusing on the prognostic proteomic features of GSRCC. Given this knowledge gap, this study aims to comprehensively characterize the proteomic landscape of GSRCC using a reliable and reproducible DIA-PCT method. This study objectives include characterizing the heterogeneity of GSRCC, performing molecular typing, identifying potential biomarkers and therapeutic targets, and providing a resource for stratified analysis of GSRCC. To achieve these goals, the investigators selected a cohort of 112 GSRCC patients from a pool of over 10,000 gastric cancer patients and conducted a proteomic analysis using the DIA-PCT method. This meticulous approach revealed four novel proteomic subtypes of GSRCC, each exhibiting unique molecular characteristics. Additionally, the investigators discovered that PRDX2 and DDX27 can serve as predictive biomarkers for GSRCC, which were further validated in an independent cohort of 75 GSRCC patients. Furthermore, the investigators paid particular attention to the MLT-GSRCC subgroup and identified three distinct proteomic clusters among MLT-GSRCC patients. Subtype 2 within this subgroup demonstrated the poorest prognosis. Through a rigorous screening process, the investigators determined potential targets for the treatment of GSRCC. In conclusion, these findings contribute to the investigators understanding of the heterogeneity of GSRCC and provide valuable resources for future clinical stratification and targeted treatment strategies.

ELIGIBILITY:
Inclusion Criteria:

* confirmed GSRCC by pathology, where GSRCC is defined as having a percentage of signet ring cell ≥ 50%
* patients with complete medical information
* patients with survival follow-up information

Exclusion Criteria:

* patients with other malignant tumors
* presence of other pathological components (e.g., neuroendocrine carcinoma and squamous cell carcinoma, etc)
* incomplete or lost case information

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: These cases had a signet ring cell content greater than 70% and had not undergone prior chemotherapy or radiotherapy
Sampling Method: Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2023-03-02 (Actual); Primary Completion 2024-06-30 (Estimated); Study Completion 2024-07-30 (Estimated)

PRIMARY OUTCOMES:
The proteome of tissue | Lc-MS/MS was used to detect the types of proteins in the samples and the relative amounts in the samples compared with Normal adjacent tissue, an average of one month
  The samples diagnosed as GSRCC by pathology were selected as the samples with signet ring cell content > 70% as judged by 2 pathologists of associate chief physician or above and without previous radiotherapy and chemotherapy. Tumor tissues and paired nat were collected from the same patient at the time of tumor resection and stored in formalin-fixed paraffin embedding (FFPE). Liquid chromatography-mass spectrometry (LC-MS) was used to detect the proteomics in the samples. The proteins in the samples were extracted, and the proteomics in the samples was detected by LC-MS. Qualitative and quantitative analysis was performed to detect the types and content of proteins in the samples.

CONTACTS AND LOCATIONS:
Locations (1):
- Cancer Hospital of the University of Chinese Academy of Sciences (Zhejiang Cancer Hospital), Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No
This study does not involve drug clinical trials but focuses on ensuring the confidentiality of patient information. To protect patient privacy, a coding system was used instead of real names when entering patient information such as names and ages. Each patient was assigned a study identification number upon enrollment. Throughout the entire study, only the main researchers in the research team have the authority to access the true personal data of patients obtained from the electronic database (such as names and ages), and it is strictly prohibited to circulate or share this information. During the publication of the research article, the main researchers in the research team will use sample coding to replace patient privacy information (such as names) to achieve de-identification. Additionally, the protection of personal information for study participants must be maintained throughout the entire research process, and it is strictly forbidden to circulate or leak such information.

REFERENCES:
- [Result] Puccini A, Poorman K, Catalano F, Seeber A, Goldberg RM, Salem ME, Shields AF, Berger MD, Battaglin F, Tokunaga R, Naseem M, Zhang W, Philip PA, Marshall JL, Korn WM, Lenz HJ. Molecular profiling of signet-ring-cell carcinoma (SRCC) from the stomach and colon reveals potential new therapeutic targets. Oncogene. 2022 Jun;41(26):3455-3460. doi: 10.1038/s41388-022-02350-6. Epub 2022 May 26. PMID 35618879
- [Result] Fan Y, Bai B, Liang Y, Ren Y, Liu Y, Zhou F, Lou X, Zi J, Hou G, Chen F, Zhao Q, Liu S. Proteomic Profiling of Gastric Signet Ring Cell Carcinoma Tissues Reveals Characteristic Changes of the Complement Cascade Pathway. Mol Cell Proteomics. 2021;20:100068. doi: 10.1016/j.mcpro.2021.100068. Epub 2021 Mar 3. PMID 33676000
- [Result] Ge S, Xia X, Ding C, Zhen B, Zhou Q, Feng J, Yuan J, Chen R, Li Y, Ge Z, Ji J, Zhang L, Wang J, Li Z, Lai Y, Hu Y, Li Y, Li Y, Gao J, Chen L, Xu J, Zhang C, Jung SY, Choi JM, Jain A, Liu M, Song L, Liu W, Guo G, Gong T, Huang Y, Qiu Y, Huang W, Shi T, Zhu W, Wang Y, He F, Shen L, Qin J. A proteomic landscape of diffuse-type gastric cancer. Nat Commun. 2018 Mar 8;9(1):1012. doi: 10.1038/s41467-018-03121-2. PMID 29520031
- [Result] Asleh K, Negri GL, Spencer Miko SE, Colborne S, Hughes CS, Wang XQ, Gao D, Gilks CB, Chia SKL, Nielsen TO, Morin GB. Proteomic analysis of archival breast cancer clinical specimens identifies biological subtypes with distinct survival outcomes. Nat Commun. 2022 Feb 16;13(1):896. doi: 10.1038/s41467-022-28524-0. PMID 35173148
- [Result] Chen J, Liu K, Luo Y, Kang M, Wang J, Chen G, Qi J, Wu W, Wang B, Han Y, Shi L, Wang K, Han X, Ma X, Liu W, Ding Y, Wang L, Liang H, Wang L, Chen J. Single-Cell Profiling of Tumor Immune Microenvironment Reveals Immune Irresponsiveness in Gastric Signet-Ring Cell Carcinoma. Gastroenterology. 2023 Jul;165(1):88-103. doi: 10.1053/j.gastro.2023.03.008. Epub 2023 Mar 14. PMID 36921674